CLINICAL TRIAL: NCT05271617
Title: VIDAS Nephroclear CCL14 : Sample Stability Study
Brief Title: VIDAS Nephroclear (NCL) CCL14 - Sample Stability
Status: Completed | Type: Observational
Sponsor: BioMérieux (Industry)
Responsible Party: Sponsor
Other Study IDs: B3166-CTPR01
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: VIDAS® NEPHROCLEAR™ CCL14 — Measurement of CCL14 in sample aliquots after being subjected to different testing conditions

SUMMARY:
This VIDAS® NEPHROCLEAR™ CCL14 (VIDAS® NCL™ CCL14) Sample Stability clinical trial is a multicenter, prospective, and qualitative study. The main study objective is to determine sample stability conditions for the VIDAS® NEPHROCLEAR™ CCL14 Test. This test is intended to be used in conjunction with clinical evaluation in ICU patients with moderate to severe (stage 2 or 3) acute kidney injury (AKI) as an aid in the risk assessment for developing persistent severe AKI (stage 3 AKI lasting ≥ 72 hours) within 48 hours of patient assessment. The VIDAS® NEPHROCLEAR™ CCL14 Test is intended to be used in patients 21 years of age or older.

DETAILED DESCRIPTION:
Product name and intended use

The VIDAS® NEPHROCLEAR™ CCL14 Test is intended to be used in conjunction with clinical evaluation in ICU patients with moderate to severe (stage 2 or 3) acute kidney injury (AKI) as an aid in the risk assessment for developing persistent severe AKI (stage 3 AKI lasting ≥ 72 hours) within 48 hours of patient assessment. The VIDAS® NEPHROCLEAR™ CCL14 Test is intended to be used in patients 21 years of age or older.

Product description

The VIDAS® NEPHROCLEAR™ CCL14 Test is an automated assay for use on the VIDAS® 3 instrument for the immunoenzymatic quantitative determination of C-C motif chemokine ligand 14 (CCL14) protein in human urine using the Enzyme Linked Fluorescent Assay (ELFA) technique.

Trial Design Overview

This VIDAS® NEPHROCLEAR™CCL14 (VIDAS® NCL™ CCL14) clinical trial is a multicenter, prospective, and qualitative study. 40 to 80 samples collected and tested from subjects enrolled in a related trial will also be tested on the VIDAS® 3 instrument and test.

Trial objectives

The objective of this trial is to identify suitable storage conditions for samples tested using the VIDAS® NCL™ CCL14 for the full measuring range of the assay (0.2 ng/mL to 30 ng/mL). To this end, samples will be tested under the following conditions:

* Fresh, and tested within approximately 2 hours of collection,
* After one freeze-thaw cycle,
* After two freeze-thaw cycles,
* After storage at ambient temperature for approximately 5 hours (tested 5 to 7 hours from collection time), and
* After storage at 2 - 8 ºC for approximately 24 hours (tested 24 to 26 hours from collection time)

Samples collected from at least 40 subjects with urine CCL14 levels spanning the assay measuring range will be analyzed among these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 21 years of age or older;
* Receiving care in an intensive care unit;
* Expected to remain in the ICU for at least 48 hours after enrollment;
* Use of indwelling urinary catheter as standard care at the time of enrollment;
* Subject must have acute kidney injury (KDIGO Stage 2 or Stage 3) at the time of sample collection;
* Urine sample must be collected within 36 hours of meeting KDIGO Stage 2 criteria;
* Written informed consent provided by patient or legally authorized representative (LAR).

Exclusion Criteria:

* Prior kidney transplantation;
* Comfort-measures-only status;
* Already receiving dialysis (either acute or chronic) or in imminent need of dialysis at the time of enrollment;
* Known infection with human immunodeficiency virus (HIV) or active hepatitis (acute or chronic); (NOTE: HIV or hepatitis testing will not be performed for enrollment in this study.)
* Special populations, pregnant women, prisoners or institutionalized individuals;

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU patients with moderate to severe (stage 2 or 3) acute kidney injury (AKI), who qualify based on the criteria described above. These participants are recruited under a separate protocol IRB approved protocol. This protocol covers testing of leftover samples only.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Sample stability conditions | one sample will be collected per participant, aliquots will be tested at various conditions: fresh, after one to two freeze-thaw cycles, after refrigeration for 24 hours and after 6 hours at room temperature
  Detection of CCL14 levels in urine, spanning the measuring range of the assay for several sample conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No